CLINICAL TRIAL: NCT05200689
Title: Post-Operative Kinesio Taping Impact on Pain in Thoracotomy vs Thoracoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Quds University (Other)
Collaborators: Makassed Hospital (Other); Assiut University (Other); Tanta University (Other); Papworth Hospital NHS Foundation Trust (Other Government); European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01/REC-CT/2021; 35070/11/21 (Other: Tanta University)
Record Dates: First submitted 2021-12-20; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Pain
Keywords: Kinesiotaping; Postoperative Pain; Thoracic Surgery; Comparative; Uniportal VATS; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thoracotomy, KT (Experimental): Patients in this group will undergo the same analgesia protocol as other groups. They will undergo the thoracotomy protocol, alongside the KT protocol.
  Interventions: Device: Kinesiotaping (KT)
- Thoracoscopy, KT (Experimental): Patients in this group will undergo the same analgesia protocol as other groups. They will undergo the thoracoscopy protocol, alongside the KT protocol.
  Interventions: Device: Kinesiotaping (KT)
- Thoracotomy, Non-KT (No Intervention): Patients in this group will undergo the same analgesia protocol as other groups. They will undergo the thoracotomy protocol, without the KT protocol.
- Thoracoscopy, Non-KT (No Intervention): Patients in this group will undergo the same analgesia protocol as other groups. They will undergo the thoracoscopy protocol, without the KT protocol.

INTERVENTIONS:
Device: Kinesiotaping (KT) — Kinesio taping will only be applied for a period of 5 days. Initial Kinesio taping will first occur one day after surgery.
  It will be placed directly on the chest wall on a trigger point. Physiotherapists will be instructed to maintain a standard Tape length (To body size ratio) and tension among all patients of all KT groups. The edges of the tape must be rounded, to prevent premature peeling. The adhesive side of the tape must not be touched after removing its backing, to prevent any decrease in tape adherence. It will be applied using both I and Star applications. Star and I KT application is done directly above the main pain trigger point. This point is found via chest palpitations. The Tape will be replaced every 48 hours by the physiotherapist until the end of therapy. The tape must be placed after stretching the skin.
  Other Names: Kinesio Tex Gold; K-active kinesiology tape
  Arms: Thoracoscopy, KT; Thoracotomy, KT

SUMMARY:
The project is of a comparative nature. It seeks to study pain reduction following two forms of chest surgery and compare results between both procedures. It will use kinesio taping as the studied pain reducer. It will involve 4 study groups, 2 per surgical procedure, and among those 2 main groups, 2 subgroups each where 1 has kinesio taping and the other doesn't.

With this, the project hopes to offer new forms of pain reduction that are more cost effective and are associated with less adverse effects. Furthermore it would decrease pain killer intake which is a contemporary challenge of medicine.

DETAILED DESCRIPTION:
Fueled by its utmost importance, thoracic surgery has quickly evolved to produce techniques that improve its means and purposes, but most importantly fully harness its goals. Thoracic surgeries include multiple techniques; thoracotomy and thoracoscopy are among the most highly applied types since they are involved in the diagnosis and treatment of lung cancer, cardiovascular disease, and other comorbidities, but most notably are the hallmark of lung resection.

Thoracotomy is surgery to open the chest. This procedure involves an incision in the thorax, between the ribs, to allow for operating on the lungs. A surgeon can use this incision to remove part of or the whole lung. Usually, this is done to treat lung cancer. Sometimes it's used to treat problems with the heart or other structures in the chest, such as the diaphragm. On the other hand, thoracoscopy is a surgical procedure for the examination of the chest, particularly the pleural cavity by means of a thoracoscope. Thoracoscopy can be done as part of the Video-Assisted Thoracic Surgery procedure (VATS). Uniportal VATS makes use of 1 single port incision.

Both thoracoscopy and thoracotomy have been thoroughly studied by recent literature, and even compared. However, when properly surveyed, research is found to be lacking in the field of morbidity reduction, namely when concerning pain management. This is quite alarming as the main complication of thoracic surgeries is pain, which may even extend to post-thoracotomy pain syndrome (PTPS), which occurs in 21 to 61% of patients and may persist up to four to five years after surgery in 30% of patients.

As pain is a major debilitating factor to the patient, decreasing it will serve as a major improvement for patient morbidity and satisfaction.

Analgesics are still considered one of the most effective approaches in terms of pain relief. Though the use of analgesics has been recently viewed to approach the limits of abuse, both economically and pharmacologically. This includes the epidemic overuse of opioids and such. This issue has also been at the forefront of recent medical research and at the top of the medical world's agenda for the past few years. This calls the scientific community to find a proper solution.

Although new techniques for postsurgical pain management are emerging currently, especially for thoracic surgeries, the use of these techniques is still debated. Kinesio Taping (KT) is one of those techniques. Its use has been supported in pain relief and hastens patient discharge.

This technique was introduced by Kenzo Kane, a chiropractor, in 1979 in Japan. It is an elastic bonding material containing high tensile capacity, which ensures the free movement of the application area without the need for drugs or chemicals. It is designed to mimic the skin's elasticity to allow for the use of the patients' full range of motion. Once applied to the skin, it also recoils slightly to lift the skin. This is believed to help create a microscopic space between the skin and underlying tissue.

Physical therapists have used kinesiology tape to lift the skin over tense, knotted muscles as well as to treat other disorders including rheumatic, neurological, lymphatic, and vascular disorders in recent years. Despite the lack of clarity regarding the effects of KT on pain, KT may still provide a sufficient stimulus to promote mechanisms that relieve and inhibit pain.

However, there are conflicting views and an overall lack of research regarding the effectiveness of applying Kinesio Taping in pain relief after thoracic surgeries, taking into consideration that analgesics are administered to patients after thoracic surgeries.

This research aims to check the possibility of reducing post-operative pain after thoracic surgeries and equally decrease the use of narcotics/analgesics through the application of kinesio taping.

Aims and Objective:

A. To check the possibility of reducing post-operative pain after thoracic surgeries and the use of narcotics/analgesics through applying the Kinesio tape around the surgical incision.

B. To observe the respective degree of pain reduction in thoracotomies in contrast to uniportal VATS thoracoscopies through kinesiotherapy.

Research Design and Methods:

Study Design:

This is an international multicenter clinical trial that will be conducted at Al Makassed Islamic Charitable Hospital in Jerusalem, Palestine, the Assiut University Hospital in Assiut, Egypt, the Tanta University Hospital in Tanta, Egypt, the Royal Papworth Hospital in Cambridge, the United Kingdom, and the European Institute of Oncology in Milan, Italy. The trial will be registered in clinicaltrials.gov. Registration will be sought after ethical approval, in correspondence with the associated persons.

A. Population:

The population of the study extends to thoracic surgery patients who will undergo thoracotomy and thoracoscopy in the form of uniportal VATS at the Al-Makassed Hospital department of surgery, and other associated centers, and will experience pain following their surgeries.

B. Sample:

Patients will be sampled via systematic sampling, at a rate of ⅕ for thoracoscopies and 1/1 for thoracotomies (These rates apply for Al Makassed, rates will differ per center).

C. Procedure:

Patients that fit within the project's parameters will be asked to fill out consent forms, after which initial data will be taken prior to their surgery.

The study's surgical team will also execute uniportal VATS thoracoscopies and thoracotomies in an identified operative protocol, accompanied by specific techniques for anesthesia, described as follows:

All patients will be under general anesthesia. Intraoperative single-lung ventilation will be achieved via a double-lumen tube. An arterial line will be used for hemodynamic and blood gas monitoring. Intravenous lines can be applied peripherally for drug and fluid administration. Foley catheters may be used at the surgical teams' discretion. 3-level Intercostal block (20 CC of the mixture of drugs prepared by the anesthesiologist, CC: Cubic centimeters) will be performed intraoperatively. It will involve the intercostal space where the incision will be made, as well as the space above and below.

This will apply to all patients. For patients in the uniportal VATS thoracoscopy group, they will be placed in a lateral decubitus position, with both arms along the body, otherwise known as the prayer's position. The bed for the procedure will be flexed to its fullest extent. The breakpoint will be just above the superior iliac crest. This will serve to spread the intercostal spaces. To allow for the coordination of movements between the surgeon and the assistant, they will be positioned in front of the patient and will permit them to share thoracoscopic vision throughout the whole procedure. The scrub nurse will be positioned behind the patient.

A single 3-5 cm incision will be made in the 5th intercostal space around the area of the anterior axillary line. This position will ease hilar dissection and stapler insertion. A wound protector can be used according to the surgeon's preference. To avoid the contamination of the camera, and to facilitate its insertion, the wound will be retracted via 2 stitches, 1 on each side. The thoracoscope will be inserted and maintained in the posterior part of the incision.

For patients in the thoracotomy group, they will undergo posterolateral thoracotomies. Primarily, patients will be placed in a lateral decubitus position, with padding to the elbows and joints provided. The legs must be separated, with the lower leg flexed. The lower arm will be flexed and placed next to the head, while the upper arm will be left to hang over the bed. The patients' position will be maintained by straps.

The incision will follow the course of the underlying ribs. The incision will extend from 7 cm from the mid spinal line to the anterior axillary line. This is at the level of the 6th rib. The incision will extend to dissect the latismus Dorsi muscle. Incision of the intercostal muscle is made carefully and towards the lower rib to avoid nerve damage. Rib spreading must be performed slowly and progressively.

Please note that the surgical and anaesthesia procedures are not the exposure, but instead are procedures that the participants will undergo regardless of our project, to treat their existing pathologies. The investigators are simply recruiting these individuals for KT therapy as part of the clinical trial. Standardization of the procedures is still however essential for minimizing confounders, and is done in a medically and surgically sound way.

Physiotherapy and Kinesio tape protocol:

Both KT and Non-KT groups will be exposed to the same protocol. Further patient data will then be taken throughout the period of the first 21 days following the operation, to monitor the effect of Kinesio taping. As the patient monitoring period will last for 3 weeks after the operation; there will be telephonic interviews with the patients who discharge before this period in order to evaluate their pain intensity.

Kinesio taping will only be applied for a period of 5 days. Initial Kinesio taping will first occur one day after surgery. The study will use Kinesio Tex Gold/K-active kinesiology tape and will apply it to all patients of the KT groups. Please note that the tape will be provided by the centers participating in the study. It is made from polymer elastic wrapped in cotton and is latex-free/skin adhesive cotton fabric. It is thus suitable for sensitive skin and offers breathability and is water repellent. It will be placed directly on the chest wall on a trigger point. Physiotherapists will be instructed to maintain a standard Tape length (To body size ratio) and tension among all patients of all KT groups. The edges of the tape must be rounded, to prevent premature peeling. The adhesive side of the tape must not be touched after removing its backing, to prevent any decrease in tape adherence. It will be applied using both I and Star applications, which were empirically found to decrease pain. Star and I KT application is done directly above the main pain trigger point. This point is found via chest palpitations. The Tape will be replaced every 48 hours by the physiotherapist until the end of therapy. Most importantly, the tape must be placed after stretching the skin, to allow the elastic Kinesio taping to lift the skin and provide proper space correction to the underlying soft tissue.

Per Center, the same physiotherapist will apply the tape to all patients involved in the study. The area where the tape will be applied will be clean and shaven as necessary and must be oil and lotion-free before the application. Physiotherapists must be sure that patients that were exercising beforehand have had perspiration subside prior to application. After application, patients must be instructed to abstain from activities that would lead to sweating, and avoid getting wet for an hour (Limit excess activity and avoid water). Patients will also be instructed to gently pat the tape to dry it after sweating, swimming, or showering that may occur after the 1 hour period. Due to the tape's lack of sterility, it will not be placed over wounds or bandages (this includes scrapes, cuts, burns, sunburn, and skin irritation). The tape must be rubbed to activate the acrylic glue.

Intraoperative analgesia protocol:

Furthermore, the surgical team must be the same for the thoracotomy groups and thoracoscopy groups respectively in individual centers.

All patient groups will be provided with required and demanded analgesics and narcotics postoperatively, via a unified drug protocol. The protocol is as follows:

* On postoperative days 1, 2, 3: intravenous paracetamol (1 g three times a day: at 8 am, 4 pm, and 12 pm); epidural naropin (0.2% at 4 ml per hour) and subcutaneous morphine (5 mg/day, at patient request).
* From postoperative day 4 until discharge: oral paracetamol/codeine (500/30 mg twice/day: at 6 am and 6 pm) and oral ibuprofen (600 mg twice/day: at 12 am and 12 pm).
* Supplemental analgesics [non-steroidal anti-inflammatory drugs (NSAID) and opioids] are available at patient request in both groups Patients that request further analgesia will have that data recorded for them.

D. Data collection:

Data will be collected prospectively. Data will first be collected prior to KT after patient recruitment, and then patients will be followed for 3 weeks. Data will be collected once prior to KT, and then after kinesiotherapy starts pain will be recorded, followed by another record on the third day of surgery, the seventh day of surgery, and a final assessment on the 21st day of surgery.

Data will be collected via a questionnaire. The patient's file number will be determined. A measure of pain pre-surgery and post-operatively will be made. Collected data will include demographics (age and sex), anthropometrics (weight, Height, BMI), and, smoking status (yes/No/formerly), lung cancer (the type and the stage if present), surgical approach (open thoracotomy or uniportal VATS), postoperative complications, duration of postoperative pain. Accessory analgesics will also be recorded.

The pre-operative preparation will be checked for each patient. According to the US Food and Drug Administration (FDA), some of the most important laboratory tests are going to be performed before surgery as a part to identify potential problems that might complicate surgery if not detected and treated early. These tests are:

* Chest X-rays that may help to diagnose causes of shortness of breath, chest pain, cough, fever of unknown origin, and other abnormal heart, respiratory, and lung sounds.
* Electrocardiogram (ECG or EKG).
* Urinalysis which maybe be used to diagnose kidney and bladder, it also detects drugs present in the body.
* CBC (CBC: Complete Blood Count), including White blood count since it may be used to diagnose fever of unknown origin, infection, and use of drugs known to affect white blood counts.

Pain will be measured through multiple approaches. Pain intensity will be measured via the VAS pain scales. Pain will be assessed as follows: On the postoperative day 1 (before, and after tape application), 3, 5, 7, and 21. The measurement of chest pain after surgery will be performed by patient self-assessment

• Visual Analog Scale for Pain "VAS-Pain is a unidimensional measure of pain intensity. It is a continuous, single-item scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Those descriptors are "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended. The cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm). It takes less than 1 minute to complete. The VAS is administered as a paper and pencil measure. As a result, it cannot be administered verbally or by phone. In this study, the VAS-pain scores were assessed in different settings including resting, during deep breathing, coughing, and bending to the operated side".

The VAS pain scale will be used at every point of pain measurement. A table of preoperative and postoperative lab data and postoperative complications including blood loss will be made.

Data will be collected by independent observers.

E. Clinical Significance:

The results of this study have a wide range of applicability to all patients who might undergo thoracoscopy or thoracotomy with the implementation of Kinesio taping as a form of pain and morbidity reduction therapy should the investigators prove their hypothesis, and it can fuel the search for other forms of pain reduction should they reject it. The results of the study can also be used as a basis for future research into thoracic surgery for starters and kinesiotherapy as a whole.

Overall this study will provide evidence-based practice for future guidelines concerned with the topic. It will also benefit patients who undergo these procedures by decreasing postoperative pain as well as the consumption of analgesics which is both economically and mentally favorable. It furthermore helps influence healthcare professionals to less morbid procedures between thoracotomy and thoracoscopy as a product of this comparative research.

F. Data Analysis:

Data Analysis will be done through the use of IBM SPSS (IBM: International Business Machines, SPSS: Statistical Product and Service Solutions) for Windows version 16.0.

Accordingly, the investigators will see whether the used thoracic surgery techniques and the pain relief approach will differ significantly between these groups or not.

The investigators believe that a statistically significant decrease in postoperative pain intensity, duration, and painkiller need signifies that Kinesio taping does in fact signify a decrease in post-operative pain. This data will be collected from all groups. Non-KT and KT groups of the same surgical group will be compared, and KT groups will be compared among each other.

ELIGIBILITY:
Inclusion Criteria:

* Single port VATS thoracoscopies
* Patients that undergo thoracotomy or thoracoscopy at associated centers
* Patients within the age range (18-64) years.

Exclusion Criteria:

* Preexisting conditions
* Certain surgical complication
* KT and analgesics-related contraindications
* Patients that offer logistic difficulties.
* Patients that suffer from recent chest trauma (Within 6 months), pre-existing chest pain
* Rib resection, pleuralesis, parietal pleura involvement in the surgery
* Surgeries with increased involvement of the chest, vertebrobasilar insufficiency
* Inflammatory diseases
* Neurologic diseases
* Congenital diseases
* Fractures, dislocations, infections
* Dural perforations, spinal cord damage with abscess development due to nerve block
* Patients who have contraindications to KT, especially those who suffer from DVT (DVT: Deep Vein Thrombosis), skin Pathologies, and diseases, especially relating to the chest area
* Patient with congestive heart failure
* Patients that experience skin sensitivity or allergy to the Kinesio taping
* Patients who undergo other forms of pain reduction therapy such as massages
* The lack of patient consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-01-09 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain: Change in VAS Pain Scale | 21 days
  Degree of change in postoperative pain. It will be measured 5 times. Postoperative pain will be measured via the VAS pain scale. It will also be estimated based on the patients' request for further analgesia.
  The VAS Scale stands for: Visual Analog Scale. Minimum Score: 0 Maximum Score: 100 Higher scores signify worse pain and thus a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Bael, Principal Investigator — Al-Quds University; Raya Amro, Principal Investigator — Al-Quds University; Mayar Idkedek, Principal Investigator — Al-Quds University
Locations (5):
- Egypt (2):
  - Assiut Uniersity, Asyut
  - Tanta University, Tanta
- European Institute of Oncology, Milan, Italy
- Al-Makased Hospital, East Jerusalem, Palestinian Territories
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Howington JA, Blum MG, Chang AC, Balekian AA, Murthy SC. Treatment of stage I and II non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e278S-e313S. doi: 10.1378/chest.12-2359. PMID 23649443
- [Result] Kurt Saruhan H, Toprak M. Pain-diminishing and quality of life-related outcomes of Kinesio taping in patients on non-steroidal anti-inflammatory drug therapy for post-thoracotomy pain syndrome. Turk J Phys Med Rehabil. 2020 May 18;66(2):147-153. doi: 10.5606/tftrd.2020.4068. eCollection 2020 Jun. PMID 32760891
- [Result] Alzahrani T. Pain relief following thoracic surgical procedures: A literature review of the uncommon techniques. Saudi J Anaesth. 2017 Jul-Sep;11(3):327-331. doi: 10.4103/sja.SJA_39_17. PMID 28757835
- [Result] Zeng R, Tian K, Xiao Z. Effectiveness of thoracic kinesio taping on respiratory function and muscle strength in patients with chronic obstructive pulmonary disease: A protocol of randomized, double-blind placebo-controlled trial. Medicine (Baltimore). 2021 Apr 9;100(14):e25269. doi: 10.1097/MD.0000000000025269. PMID 33832089
- [Result] Imperatori A, Grande A, Castiglioni M, Gasperini L, Faini A, Spampatti S, Nardecchia E, Terzaghi L, Dominioni L, Rotolo N. Chest pain control with kinesiology taping after lobectomy for lung cancer: initial results of a randomized placebo-controlled study. Interact Cardiovasc Thorac Surg. 2016 Aug;23(2):223-30. doi: 10.1093/icvts/ivw110. Epub 2016 Apr 29. PMID 27130717
- [Result] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Result] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Result] Laursen LO, Petersen RH, Hansen HJ, Jensen TK, Ravn J, Konge L. Video-assisted thoracoscopic surgery lobectomy for lung cancer is associated with a lower 30-day morbidity compared with lobectomy by thoracotomy. Eur J Cardiothorac Surg. 2016 Mar;49(3):870-5. doi: 10.1093/ejcts/ezv205. Epub 2015 Jun 18. PMID 26088592
- [Result] Luz Junior MA, Sousa MV, Neves LA, Cezar AA, Costa LO. Kinesio Taping(R) is not better than placebo in reducing pain and disability in patients with chronic non-specific low back pain: a randomized controlled trial. Braz J Phys Ther. 2015 Nov-Dec;19(6):482-90. doi: 10.1590/bjpt-rbf.2014.0128. Epub 2015 Oct 9. PMID 26647750
- [Result] Ristow O, Pautke C, Victoria Kehl, Koerdt S, Schwarzler K, Hahnefeld L, Hohlweg-Majert B. Influence of kinesiologic tape on postoperative swelling, pain and trismus after zygomatico-orbital fractures. J Craniomaxillofac Surg. 2014 Jul;42(5):469-76. doi: 10.1016/j.jcms.2013.05.043. Epub 2013 Jul 4. PMID 23830769
- [Result] Laborie M, Klouche S, Herman S, Gerometta A, Lefevre N, Bohu Y. Inefficacy of Kinesio-Taping((R)) on early postoperative pain after ACL reconstruction: Prospective comparative study. Orthop Traumatol Surg Res. 2015 Dec;101(8):963-7. doi: 10.1016/j.otsr.2015.09.025. Epub 2015 Nov 14. PMID 26589192
- [Result] Parreira Pdo C, Costa Lda C, Hespanhol LC Jr, Lopes AD, Costa LO. Current evidence does not support the use of Kinesio Taping in clinical practice: a systematic review. J Physiother. 2014 Mar;60(1):31-9. doi: 10.1016/j.jphys.2013.12.008. Epub 2014 Apr 24. PMID 24856938
- [Result] Elabd AM, Ibrahim AR, Elhafez HM, Hussien HA, Elabd OM. Efficacy of Kinesio Taping and Postural Correction Exercises on Levator Scapula Electromyographic Activities in Mechanical Cervical Dysfunction: A Randomized Blinded Clinical Trial. J Manipulative Physiol Ther. 2020 Jul-Aug;43(6):588-596. doi: 10.1016/j.jmpt.2019.05.010. Epub 2020 Jul 21. PMID 32709516
- [Result] Krajczy M, Bogacz K, Luniewski J, Szczegielniak J. The influence of Kinesio Taping on the effects of physiotherapy in patients after laparoscopic cholecystectomy. ScientificWorldJournal. 2012;2012:948282. doi: 10.1100/2012/948282. Epub 2012 May 3. PMID 22645478
- [Result] Ulu M, Gozluklu O, Kaya C, Unal N, Akcay H. Three-Dimensional Evaluation of the Effects of Kinesio Taping on Postoperative Swelling and Pain after Surgically Assisted Rapid Palatal Expansion. J Oral Maxillofac Res. 2018 Dec 30;9(4):e3. doi: 10.5037/jomr.2018.9403. eCollection 2018 Oct-Dec. PMID 30746052
- [Result] Chan MC, Wee JW, Lim MH. Does Kinesiology Taping Improve the Early Postoperative Outcomes in Anterior Cruciate Ligament Reconstruction? A Randomized Controlled Study. Clin J Sport Med. 2017 May;27(3):260-265. doi: 10.1097/JSM.0000000000000345. PMID 27428680
- [Result] Brockmann R, Klein HM. Pain-diminishing effects of Kinesio(R) taping after median sternotomy. Physiother Theory Pract. 2018 Jun;34(6):433-441. doi: 10.1080/09593985.2017.1422205. Epub 2018 Jan 8. PMID 29308962
- [Result] Nobel TB, Adusumilli PS, Molena D. Opioid use and abuse following video-assisted thoracic surgery (VATS) or thoracotomy lung cancer surgery. Transl Lung Cancer Res. 2019 Dec;8(Suppl 4):S373-S377. doi: 10.21037/tlcr.2019.05.14. No abstract available. PMID 32038918
- [Result] Joshi GP, Bonnet F, Shah R, Wilkinson RC, Camu F, Fischer B, Neugebauer EA, Rawal N, Schug SA, Simanski C, Kehlet H. A systematic review of randomized trials evaluating regional techniques for postthoracotomy analgesia. Anesth Analg. 2008 Sep;107(3):1026-40. doi: 10.1213/01.ane.0000333274.63501.ff. PMID 18713924
- [Result] Guner S, Alsancak S, Koz M. Effect of two different kinesio taping techniques on knee kinematics and kinetics in young females. J Phys Ther Sci. 2015 Oct;27(10):3093-6. doi: 10.1589/jpts.27.3093. Epub 2015 Oct 30. PMID 26644651
- [Result] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Result] Joyce CR, Zutshi DW, Hrubes V, Mason RM. Comparison of fixed interval and visual analogue scales for rating chronic pain. Eur J Clin Pharmacol. 1975 Aug 14;8(6):415-20. doi: 10.1007/BF00562315. PMID 1233242
- See also: Related Info — https://www.healthline.com/health/thoracotomy
- See also: Related Info — https://www.cancer.org/treatment/understanding-your-diagnosis/tests/endoscopy/thoracoscopy.html
- See also: Related Info — https://www.healthline.com/health/kinesiology-tape
- See also: Related Info — https://stanfordhealthcare.org/medical-treatments/g/general-surgery/procedures/surgery-preparation.html